A phase II study of Platinum-doublet chemotherapy in combination with nivolumab as first-line treatment, in subjects with unresectable, locally advanced or metastatic G3
Neuroendocrine Neoplasms (NENs) of the gastroenteropancreatic (GEP) tract or of unknown (UK) origin. (GETNE T1913).

## **NICE-NEC STUDY**

## **FINAL STATISTICAL REPORT (2022)**

9th of November 2022





#### 1. TABLE OF CONTENTS 2. PATIENTS RECRUITED AND STUDY POPULATIONS 5 2.1. SCREENING FAILURES 5 2.2. PATIENT POPULATIONS 6 RESULTS 8 3.1. EVALUABLE PATIENTS 8 3.2. **BASELINE CHARACTERISTICS** 9 3.2.1. BASELINE - DEMOGRAPHIC DATA 9 3.2.2. BASELINE - CANCER HISTORY 11 3.3. **BASELINE - ANALYTICS** 15 3.4. 15 Baseline - Hematology and Coagulation 17 3.5. Baseline - Biochemistry, Thyroid Function and Serology 22 36 Baseline - Other Determinations 4. Treatment exposure 24 24 4.1. Induction Phase 4.2. Maintenance Phase 29 4.3. Total duration of treatment with Nivolumab 35 4.4. Cycles administered after progression 35 END OF TREATMENT - END OF STUDY - FOLLOW-UP 4.5. 36 4.5.1. End of treatment 36 4.5.2. End of Study 36 37 4.5.3. Follow-up (all patients) 4.5.4. Follow-up (only alive patients) 37 4.6. PRIMARY ENDPOINT: OVERALL SUVIVAL (OS) 38 4.7. SECONDARY ENDPOINTS 40 4.7.1. PROGRESSION FREE SURVIVAL (PFS) 40 40 4.7.2. Events: Progressions/Deaths 4.7.3. ORR: Objective Response Rate 42 42 4.7.4. Best Overall Response 4.7.5. Duration of Response 42 43 4.7.5.1. Figure: Waterfall plot. Maximum % total change with BOR 4.7.5.2 Figure: Waterfall plot. Maximum % total change VS BOR 44

| 4.7.5.3 Figure: Waterfall plot. Maximum % total change VS pRIMARY LOCATION | 45 |
|---|---|
| 4.7.5.4 Figure: Waterfall plot. Maximum % total change VS KI67 | 46 |
| 4.7.5.4 Figure: Waterfall plot. Maximum % total change VS DIFFERENTATION TUMOUR | 47 |
| 4.7.5.2. Figure: Spider plot. Maximum % total change | 48 |
| 4.7.5.5 Figure: Spider plot. Maximum % total change VS | |
| DIFFERENTIATION | 49 |
| 4.7.5.6 Figure: Spider plot. Maximum % total change VS BOR | 50 |
| 4.7.5.7 Figure: Spider plot. Maximum % total change VS CGA | 51 |
| 4.7.5.8 Figure: Spider plot. Maximum % total change VS NSE | 52 |
| 4.8. OS STRATIFIED BY FACTORS OF INTEREST: DIFFERENTIATED/ K<br>PRIMARY TUMOUR LOCATION / CGA / NSE | i67/<br>53 |
| 4.8.1. OS vs Differentiation | 53 |
| 4.8.1.1. Figure: OS vs Differentiation. Kaplan Meier graph | 54 |
| 4.8.2. OS vs Ki67 | 55 |
| 4.8.2.1. Figure: OS vs Ki67. Kaplan Meier graph | 56 |
| 4.8.3. OS vs Location | 57 |
| 4.8.3.1. Figure: OS vs Location. Kaplan Meier graph | 58 |
| 4.8.4. OS vs CGA | 59 |
| 4.8.4.1. Figure: OS vs CGA Kaplan Meier graph | 60 |
| 4.8.5. OS vs NSE | 61 |
| 4.8.5.1. Figure: OS vs NSE Kaplan Meier graph | 62 |
| 4.9. PFS STRATIFIED BY FACTORS OF INTEREST: DIFFERENTIATED/<br>Ki67/ PRIMARY TUMOUR LOCATION / CGA / ENOLASE | 63 |
| 4.9.1. PFS vs Differentiation | 63 |
| 4.9.1.1. Figure: PFS vs Differentiation. Kaplan Meier graph | 64 |
| 4.9.2. PFS vs Ki67 | 65 |
| 4.9.2.1. Figure: PFS vs Ki67. Kaplan Meier graph | 66 |
| 4.9.3. PFS vs Location | 67 |
| 4.9.3.1. Figure: PFS vs Location. Kaplan Meier graph | 68 |
| 4.9.4. PFS vs CGA | 69 |
| 4.9.4.1. PFS vs CGA (2) | 69 |
| 4.9.4.2. Figure: PFS vs CGA Kaplan Meier graph (2) | 70 |
| 4.9.4.3. PFS vs CGA (3) | 71 |
| 4.9.4.4. Figure: PFS vs CGA Kaplan Meier graph (3) Page 3 of 83 | 72 |

| | | 4.9.4.5. | PFS vs CGA (5) | 73 |
|---|---|---|---|---|
| | | 4.9.4.6. | Figure: PFS vs CGA Kaplan Meier graph (5) | 74 |
| | 4.9 | 9.5. PF | S vs Enolase | 75 |
| | | 4.9.5.1. | Figure: PFS vs NSE Kaplan Meier graph | 76 |
| | 4.10<br>Ki67 | _ | STRATIFIED BY FACTORS OF INTEREST: DIFFERENTIATE<br>RY TUMOUR LOCATION / CGA / NSE | ED/<br>77 |
| | 4. | 10.1. N | MULTIVARIATE ANALYSIS OF PFS AND OS | 81 |
| | | 4.10.1.1. | Factors included in the multivariate analysis of the PFS (1) | 81 |
| | | 4.10.1.2. | Factors included in the multivariate analysis of the PFS (2) | 85 |
| | | 4.10.1.3. | Factors included in the multivariate analysis of the OS (1) | 89 |
| | | 4.10.1.4. | Factors included in the multivariate analysis of the OS (2) | 94 |
| 5. | . Sa | afety anal | ysis | 99 |
| | 5.1. | Inducti | on | 100 |
| | 5.2. | Mainte | nance | 110 |
| | 5.3. | Genera | al | 115 |

**NICE-NEC** a phase II study of Platinum-doublet chemotherapy in combination with nivolumab as first-line treatment, in subjects with unresectable, locally advanced or metastatic G3 Neuroendocrine Neoplasms (NENs) of the gastroenteropancreatic (GEP) tract or of unknown (UK) origin. (GETNE T1913).

Primary endpoint is 12 m OS.

Secondary endpoints include ORR, and PFS by RECIST 1.1 and safety.

The database for the results of the following report was locked down on the XX<sup>th</sup> of XX 202X.

# 2. PATIENTS RECRUITED AND STUDY POPULATIONS

## 2.1. SCREENING FAILURES

Table 2: List of patients: screening Failure Reasons

| Patient number Screening failure | Reason Screening failure |
|----------------------------------|--------------------------|

#### 2.2. PATIENT POPULATIONS

#### **Enrolled**

All participants who signed informed consent and were registered.

Table 3: Enrolled population

| | Overall (N=) |
|----------|--------------|
| Enrolled | |
| Yes | |
| No | |

#### **Treated**

All participants who received at least one dose of any study medication. This is the primary dataset for dosing and safety analysis.

Table 4: Treated population

| | Overall (N=) |
|---------|--------------|
| Treated | |
| Yes | |
| No | |

Table 5: Treated population: Reason excluded

#### Response-Evaluable

All treated subjects who have a baseline and at least one on-treatment imaging evaluation or had progression or death prior to the first on-treatment scan.

#### **REASON FOR EVALUATION**

Table 6: Response-Evaluable population

| | Overall (N=) |
|-----------------------------|--------------|
| Response-Evaluable analysis | |
| set | |
| Yes | |
| No | |

Table 7: Response-Evaluable population: Reason excluded

| Patient<br>number | Response-<br>Evaluable<br>population | Response<br>reason | 1st Tumor<br>assessment<br>measurement<br>(lesions) | PD<br>dat<br>e | First<br>FU | EOS<br>reason | EO<br>S<br>date | First<br>treatment<br>admin |
|---|---|---|---|---|---|---|---|---|

#### 3. RESULTS

The database for the results of the following report was locked down on the XX<sup>th</sup> of XXX 202X.

#### 3.1. EVALUABLE PATIENTS

Regarding the efficacy analysis the *Response-Evaluable* population will be used (n=).

Table 8: Populations and Hospital

| Overall | Overall (N=) |
|----------------------------------------------------|--------------|
| Enrolled | |
| Yes | |
| No | |
| Treated | |
| Yes | |
| No | |
| Response-Evaluable analysis set | |
| Yes | |
| No | |
| Hospital | |
| CENTRO ONCOLÓGICO MD ANDERSON INTERNATIONAL ESPAÑA | |
| HOSPITAL RAMÓN Y CAJAL | |
| HOSPITAL UNIVERSITARI VALL D'HEBRON(*) | |
| HOSPITAL UNIVERSITARIO 12 DE OCTUBRE | |
| HOSPITAL UNIVERSITARIO CENTRAL DE ASTURIAS | |
| HOSPITAL UNIVERSITARIO LA PAZ | |
| HOSPITAL UNIVERSITARIO MIGUEL SERVET | |
| HOSPITAL VIRGEN DE LA VICTORIA | |
| HOSPITAL VIRGEN DEL ROCÍO | |
| INSTITUT CATALÀ D'ONCOLOGIA L'HOSPITALET (ICO) | |

## 3.2. BASELINE CHARACTERISTICS

#### 3.2.1.BASELINE - DEMOGRAPHIC DATA

Table 9: Baseline - Demographic Data

| Overall | Overall (N=) |
|----------------------------|----------------|
| Gender | O vorum (i v ) |
| Female | |
| Male | |
| Age at registration (year) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Race | |
| Caucasian | |
| Latin | |
| Unknown | |
| Weight (Kg) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Height (cm) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Systolic Blood Pressure | |
| (mmHg) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Diastolic Blood Pressure | |
| (mmHg) | |
| N<br>Maria (050/ 01) | |
| Mean (95%CI) | |
| SD<br>Madian (05% CI) | |
| Median (95%CI) | |
| Range | |
| Temperature (°C) | |
| N<br>Moon (05% CI) | |
| Mean (95%CI) | |
| SD<br>Madian (05% CI) | |
| Median (95%CI) | |

| Overall | Overall (N=) |
|------------------------------|--------------|
| Range | |
| Respiratory rate (bpm) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Pulse Rate (bpm) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| ECOG | |
| 0 | |
| 1 | |
| 2 | |
| Physical examination | |
| Normal | |
| Clinically relevant findings | |

#### 3.2.2.BASELINE - CANCER HISTORY

Table 10: Baseline - Cancer History (I)

| Overall | Overall (N=) |
|-----------------------------------|--------------|
| Cancer Type | Overall (IV) |
| Gastroenteropancreatic tract | |
| Primary Unknown | |
| Primary location | |
| Esophagus | |
| Gastric | |
| Pancreas | |
| Right colon | |
| Left colon | |
| Rectum | |
| Duodenum | |
| lleum | |
| Prostate | |
| Inguinal | |
| Unknown | |
| Primary location (grouped) | |
| Duodenum/lleum | |
| Esophagus/Gastric | |
| Pancreas | |
| Colon/Rectum | |
| Not specified/Others | |
| Primary location (Colon/Rectum vs | |
| Others) | |
| Colon/Rectum | |
| Others | |
| Initial T Stage | |
| TO To | |
| T1 | |
| T2 | |
| T3 | |
| Tx | |
| Initial N Stage | |
| N0 | |
| N1 | |
| N2 | |
| Nx | |
| Initial M Stage | |
| M0 | |
| M1 | |
| Cancer Stage at diagnosis | |
| III | |
| IV | |
| Histological grade | |
| 3 | |
| Ki-67 Index | |
| N N | |
| IN | |

| Overall | Overall (N=) |
|-----------------------|--------------|
| Mean (95%CI) | _ |
| SD | |
| Median (95%CI) | |
| Range | |
| Ki-67 categorised | |
| <=20 | |
| >20 | |
| Ki-67 categorised | |
| <=50 | |
| >50 | |
| Ki-67 categorised | |
| <=55 | |
| >55 | |
| Mitotic Rate | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Differentiation | |
| Well differentiated | |
| Poorly differentiated | |
| Functional status | |
| Functioning | |
| Non-functioning | |
| Unknown | |

Table 11: Baseline - Cancer History (II)

| Overall | Overall (N=) |
|-------------------------------------------------------------|--------------|
| Primary surgery | |
| Yes | |
| No | |
| Unknown | |
| Time since Primary surgery to treatment initiation (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Primary Surgery Outcome | |
| Missing data | |
| R0 | |
| R2 | |
| UK | |
| Radiotherapy | |
| Yes | |
| No | |
| Other cancer history | |
| Yes | |

| Overall | Overall (N=) |
|------------------------------|--------------|
| No | |
| Unknown | |
| Other cancer history specify | |
| NA | |
| Breast | |
| Colorectal adenoma | |
| Prostate adenocarcinoma | |

Table 12: Baseline - Current NEN

| Overall | Overall (N=) |
|-------------------|--------------|
| Current NEN T | |
| Stage | |
| T0 | |
| T1 | |
| T2 | |
| T3 | |
| T4 | |
| Tx | |
| Current NEN N | |
| Stage | |
| N0 | |
| N1 | |
| N2 | |
| Nx | |
| Current NEN M | |
| Stage | |
| M0 | |
| M1 | |
| Current NEN Stage | |
| III | |
| IV | |

Table 13: Baseline - Metastatic disease location

| Overall | Overall (N=) |
|---------------------------|--------------|
| Affected Organ Liver | |
| No | |
| Yes | |
| Affected Organ Lung | |
| No | |
| Yes | |
| Affected Organ Nodules | |
| No | |
| Yes | |
| Affected Organ Peritoneal | |
| No | |
| Yes | |
| Affected Organ Bone | |

| O !! | 0 " " " \ |
|----------------------------|--------------|
| Overall | Overall (N=) |
| No No | |
| Yes | |
| Affected Organ Spleen | |
| No | |
| Yes | |
| Affected Organ Soft tissue | |
| No | |
| Yes | |
| Affected Organ Others | |
| No | |
| Yes | |
| Affected Organs Number | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Affected Organs Number | |
| (categorised) | |
| 1 Organ | |
| 2 Organs | |
| 3 Organs | |
| 4 Organs | |
| 5 Organs | |
| 6 Organs | |

## 3.3. BASELINE - ANALYTICS

#### 3.4. BASELINE - HEMATOLOGY AND COAGULATION

Table 14: Baseline - Hematology and Coagulation

| Overall | Overall (N=) |
|------------------------|--------------|
| PTT Value | , |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Basophils (x 10e9/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Eosinophils (x 10e9/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Hematocrit (%) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Hemoglobine (g/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| INR Value | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Lymphocytes (x 10e9/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Monocytes (x 10e3/µL) | |
| N | |
| Mean (95%CI) | |
| Mean (307001) | |

| Overall | Overall (N=) |
|--------------------------------|---------------|
| SD | Overall (IV-) |
| Median (95%CI) | |
| Range | |
| Neutrophils (x 10e3/µL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Platelets (x 10e9/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| PT Value | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Red Blood Count (10e6/μL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| White Blood Count<br>(10e3/µL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

## 3.5. Baseline - Biochemistry, Thyroid Function and Serology

Table 15: Baseline - Biochemistry, Thyroid Function and Serology

| Overall | Overall (N=) |
|-----------------|--------------|
| Albumin (g/L) | everal (iv ) |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| ALT (U/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Amylase (U/L) | |
| N (2.73/ CV) | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| AST (U/L) | |
| <u>N</u> | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| BUN (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| CGA (ng/mL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| CGA <> 2 x ULN | |
| Missing data | |
| CGA >= 2*ULN | |
| CGA < 2*ULN | |
| Calcium (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Nange | |

| Overall | Overall (N=) |
|----------------------------|---------------|
| Creatinine Kinase (U/L) | Overall (IV-) |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Creatinine (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Direct Bilirubin (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| , , | |
| Range<br>Free T3 (pmol/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| , , | |
| Range<br>Free T4 (ng/dL) | |
| N N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| GGT (U/L) | |
| N<br>Marrie (050/ OI) | |
| Mean (95%CI) | |
| SD<br>Madian (050(CI) | |
| Median (95%CI) | |
| Range | |
| Glucose (mg/dL) | |
| N<br>Marrie (050/ OI) | |
| Mean (95%CI) | |
| SD<br>Marting (050) CD | |
| Median (95%CI) | |
| Range | |
| Indirect Bilirubin (mg/dL) | |
| N<br>Marrie (05% OI) | |
| Mean (95%CI) | |
| SD (050( O)) | |
| Median (95%CI) | |
| Range | |
| IFNy (ng/mL) | |
| N (0.52 (.01) | |
| Mean (95%CI) | |

| Overall | Overall (N=) |
|-------------------------|--------------|
| SD | |
| Median (95%CI) | |
| Range | |
| IL1 (pg/mL) | |
| N | |
| Mean | |
| SD | |
| Median | |
| Range | |
| IL6 (pg/mL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| LDH (U/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Lipase (U/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Magnesium (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Neuron-Specific Enolase | |
| (ng/mL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| NSE catgorised >2 x ULN | |
| Missing data | |
| NSE >= 2*ULN | |
| NSE < 2*ULN | |
| Phosphorus (mg/dL) | |
| N<br>M (05%(Q)) | |
| Mean (95%CI) | |
| SD (STOCK) | |
| Median (95%CI) | |
| Range | |
| Phosphatase (U/L) | |
| N | |

| 0 " | O " (A) \ |
|-------------------------|--------------|
| Overall | Overall (N=) |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Potassium (mmol/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Sodium (mmol/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| TNF-α Value | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Total Bilirubin (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Total Protein (g/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| TSH (mUI/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Urea (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Uric Acid (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| | • |

| Overall | Overall (N=) |
|---------|--------------|
| Range | |

## 3.6. BASELINE - OTHER DETERMINATIONS

Table 16: Baseline - Other Determinations

| Overall | Overall (N=) |
|---------------------------|--------------|
| Protein | <b>.</b> |
| Negative | |
| +1 | |
| Traces | |
| +2 | |
| +3 | |
| Unknown | |
| Bilirubin | |
| Negative | |
| Positive | |
| Unknown | |
| ND | |
| Blood | |
| Negative | |
| Positive | |
| Unknown | |
| ND | |
| Color/appearence | |
| Normal | |
| Abnormal | |
| ND | |
| Unknown | |
| Glucose | |
| Normal | |
| Abnormal | |
| Unknown | |
| Leukocytes esterase | |
| Negative | |
| Positive | |
| ND | |
| Unknown | |
| Nitrite | |
| Negative | |
| Positive | |
| Unknown | |
| Urobilinogen | |
| Negative | |
| Positive | |
| ND<br>Links and | |
| Unknown | |
| Ketones | |
| Negative | |
| Positive | |
| Unknown Uring Anglysis nu | |
| Urine Analysis pH<br>N | |
| Mean (95%CI) | |

| Overall | Overall (N=) |
|------------------------------|--------------|
| SD | |
| Median (95%CI) | |
| Range | |
| Urine Analysis Specific | |
| gravity | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| ECG | |
| Normal | |
| Clinically relevant findings | |
| Unknown | |
| Ecg QTc Value | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

## 4. TREATMENT EXPOSURE

Table 17: Patients in each phase

| Overall | Overall (N=) |
|--------------------------|--------------|
| Starting Induction Phase | |
| No | |
| Yes | |
| Starting Maintenance | |
| Phase | |
| No | |
| Yes | · |

#### 4.1. INDUCTION PHASE

Table 18: Adherence to Carboplatin, Etoposide and Nivolumab (Induction Phase)

| | Carboplatin (N=) | Etoposide (N=) | Nivolumab (N=) |
|---|---|---|---|
| Time duration of in induction (months) | , , , | / | , / |
| N | | | |
| Mean (95%CI) | | | |
| SD | | | |
| Median (95%CI) | | | |
| Range | | | |
| Number of cycles administered (Induction | | | |
| phase) | | | |
| 0 | | | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4<br>5 | | | |
| 5<br>6 | | | |
| Number of cycles administered (Induction | | | |
| phase) | | | |
| N | | | |
| Mean (95%CI) | | | |
| SD , | | | |
| Median (95%CI) | | | |
| Range | | | |
| Omission (Induction phase) | | | |
| Yes | | | |
| No | | | |
| Omissions number (Induction phase) | | | |
| N<br>(GTO) D | | | |
| Mean (95%CI) | | | |
| SD<br>Maria (250/20) | | | |
| Median (95%CI) | | | |



Table 19: Delay time Carboplatin (Induction Phase)

| Patient | delay time - | delay time - | delay time - | | delay time - | | | Carboplatin total delay time - |
|---|---|---|---|---|---|---|---|---|
| Number | phase C2<br>(days) | phase C3<br>(days) | phase C4<br>(days) | phase C5<br>(days) | phase C6<br>(days) | phase C7<br>(days) | phase C8<br>(days) | Induction phase(days) |

Table 20: Delay time Etoposide (Induction Phase)

| Patient<br>Number | delay time - | Etoposide<br>delay time -<br>Induction<br>phase C3<br>(days) | Etoposide<br>total delay<br>time -<br>Induction<br>phase(days |
|---|---|---|---|

Table 21: Delay time Nivolumab (Induction Phase)

| | Nivolumab | Nivolumab | Nivolumab | Nivolumab | Nivolumab | Nivolumab | Nivolumab | Nivolumab |
|---|---|---|---|---|---|---|---|---|
| Patient | delay time - | delay time - | delay time - | delay time - | delay time - | delay time - | delay time - | total delay |
| Number | landaration | Induction | Induction | Induction | Induction | Induction | Induction | time - |
| Number | phase C2 | phase C3 | phase C4 | phase C5 | phase C6 | phase C7 | phase C8 | Induction |
| | (days) | (days) | (days) | (days) | (days) | (days) | (days) | phase(days) |

## 4.2. MAINTENANCE PHASE

The following results are analyzed only in patients that started the maintenance phase.

Table 22: Adherence to Nivolumab (Maintenance Phase)

| Overall | Overall (N=) |
|-------------------------------------------------------------|--------------|
| Time duration of Nivolumab in Maintenance (months) | , , |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Nivolumab number of cycles administered (Maintenance phase) | |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| 7 | |
| 8 | |
| 9 | |
| 10 | |
| 11 | |
| 12 | |
| 13 | |
| 14 | |
| 15 | |
| 16 | |
| 17 | |
| 18 | |
| 19 | |
| 20 | |
| 21 | |
| 22 | |
| 23 | |
| 24 | |
| 25 | |
| 26 | |
| 27 | |
| Nivolumab number of cycles administered (Maintenance phase) | |
| N | |
| Mean (95%CI) | |
| SD (STACE) | |
| Median (95%CI) | |
| Range | |
| Nivolumab omission (Maintenance phase) | |
| No | |
| Yes | |

| Overall | Overall (N=) |
|------------------------------------------------|--------------|
| Nivolumab omissions number (Maintenance phase) | |
| 0 | |
| 1 | |
| Nivolumab omissions number (Maintenance phase) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Nivolumab delay (Maintenance phase) | |
| No | |
| Yes | |
| Nivolumab delay number (Maintenance phase) | |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| Nivolumab delay number (Maintenance phase) | |
| N (0.50/ OI) | |
| Mean (95%CI) | |
| SD (SECOND) | |
| Median (95%CI) | |
| Range | |

Table 23: Delay time Nivolumab (Maintenance Phase)

| Patient | | | | | | | | | | Nivoli | umab d | delay ti | me – M | lainten | ance p | hase | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | C2 C3<br>(days) (days) | C4<br>(days) | C5<br>(days) | C6<br>(days) | C7<br>(days) | C8<br>(days) | C9<br>(days) | C10<br>(days) | C11<br>(days) | C12<br>(days) | C13<br>(days) | C14<br>(days) | C15<br>(days) | C16<br>(days) | C17<br>(days) | C18<br>(days) | C19<br>(days) | C20<br>(days) | C21<br>(days) | C22<br>(days) | C23<br>(days) | C24<br>(days) | C25<br>(days) | C26<br>(days) | (da<br>s) ys) |

Table 24: List of administered dates Nivolumab (Maitenance Phase)

| Patient<br>Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | 27 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

#### 4.3. Total duration of treatment with Nivolumab

| Overall | Overall (N=) |
|-------------------------------------------------------------|--------------|
| Time duration of Nivolumab Induction + Maintenance (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

## 4.4. CYCLES ADMINISTERED AFTER PROGRESSION

Table 25: Cycles administered after progression

| | Nivolumab (N=) |
|---|---|
| Cycles after progression Nivolumab (Maintenance phase) | |
| Yes | |
| No | |
| Number of cycles after progression Nivolumab (Maintenance phase) | |
| 0 | |
| 1 | |
| 2 | |
| Number of cycles after progression Nivolumab (Maintenance phase) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

## 4.5. END OF TREATMENT - END OF STUDY - FOLLOW-UP

#### 4.5.1. END OF TREATMENT

Table 26: End of Treatment reasons

| Overall | Overall (N=) |
|-----------------------------------|--------------|
| Reason for End Of Treatment | |
| Progression | |
| Unnacceptable toxicity | |
| Investigator decision | |
| Study treatment completion | |
| Other | |
| Other reason for End Of Treatment | |
| specified | |
| Clinical impairment and death | |
| Death | |
| Esophageal mucositis | |
| Not applicable | |
| Not specified | |

#### **4.5.2. END OF STUDY**

Table 27: End of Study reasons

| Overall | Overall (N=) |
|-------------------------------|--------------|
| Reason for End Of Study | |
| Lost of follow-up | |
| Exitus | |
| Others | |
| Other reason for End Of Study | |
| specified | |
| End of study | |
| Not applicable | |

## 4.5.3. FOLLOW-UP (ALL PATIENTS)

Table 28: Median follow-up (all patients)

| Overall | Overall (N=) |
|-------------------------------------------------------|--------------|
| Time since treatment started (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Time since treatment started (months) [> 24 months of | |
| follow-up] | |
| N N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

## 4.5.4. FOLLOW-UP (ONLY ALIVE PATIENTS)

Table 29: Median follow-up (only alive patients)

| Overall | Overall (N=) |
|-------------------------------------------------------|--------------|
| Time since treatment started (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Time since treatment started (months) [> 24 months of | |
| follow-up] | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

The efficacy analyses are reported in those patients belonging to the response population as defined previously (n=).

#### 4.6. PRIMARY ENDPOINT: OVERALL SURVIVAL (OS)

As specified in the protocol the **Primary endpoint is one year OS rate** with nivolumab plus chemotherapy. This is defined as the proportion of patients that remain alive at 12 months since the beginning of treatment. OS will be censored on the last date a participant was known to be alive.

Table 30: Events type OS

| os | N | % | 95%CI |
|-------|---|---|-------|
| Alive | | | |
| Death | | | |
| Total | | | |

| Reason of death | N | % | 95%CI |
|------------------------|---|---|-------|
| Clinical deterioration | | | |
| Clinical worsening. | | | |
| Not applicable | | | |
| Progression disease | | | |
| Sepsis | | | |
| Unknown | | | |
| Total | | | |

Table 31: Median/mean OS (estimated by Kaplan-Meier)

| | Median (months) | CI 95% | Mean | CI 95% |
|------------------|-----------------|--------|------|--------|
| Overall survival | | | | |

Table 32: OS estimated survival ratio

| os | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| At 6 months | | | | |
| At 12 months | | | | |
| At 18 months | | | | |
| At 24 months | | | | |
| At 30 months | | | | |
| At 36 months | | | | |

Figure 1: Overall survival
# 4.7. SECONDARY ENDPOINTS 4.7.1.PROGRESSION FREE SURVIVAL (PFS)

As specified in the protocol **PFS** is defined as the time from the enrollment date to the date of the first documented tumor progression per RECIST 1.1, or death due to any cause. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments will be censored on the beginning of treatment date. PFS curves, PFS medians with 95% CIs, and PFS rates at 6, 12, 18, 24, 36, and 48 months with 95% CIs will be estimated using Kaplan-Meier methodology if follow-up requirements are met.

#### 4.7.2. EVENTS: PROGRESSIONS/DEATHS

Table 33: Events type PFS

| PFS (PD REcist 1.1 or Death) | N | % | 95%CI |
|------------------------------|---|---|-------|
| No | | | |
| PD (Recist 1.1) | | | |
| Death (without previous PD) | | | |
| Total | | | |

Table 34: Median/mean PFS (estimated by Kaplan-Meier)

| | Median (months) | CI 95% | Mean | CI 95% |
|---------------------------|-----------------|--------|------|--------|
| Progression free survival | | | | |

Table 35: PFS estimated survival ratio

| PFS | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| | | | | _ |
| At 6 months | | | | |
| At 12 months | | | | |
| At 18 months | | | | |
| At 24 months | | | | |
| At 30 months | | | | |
| At 36 months | | | | |

Figure 2: Progression free survival

#### 4.7.3. ORR: OBJECTIVE RESPONSE RATE

**BOR** and **ORR** are determined based on RECIST 1.1.

#### 4.7.4. BEST OVERALL RESPONSE

Table 36: ORR

| Overall Response Rate | N | % | 95%CI |
|-----------------------|---|---|-------|
| PR | | | |
| SD | | | |
| PD | | | |
| NE | | | |
| Total | | | |

Table 37: BOR: Best Overall Response

| Overall | Overall (N=) |
|--------------|--------------|
| Best Overall | |
| Response | |
| PR | |
| SD | |
| PD | |
| NE | |

<sup>&</sup>lt;sup>+</sup> The X patients with **NE** had XXX

#### 4.7.5. DURATION OF RESPONSE

The duration of response is calculated in those patients with Best Response CR or PR.

Table 38: BOR: Best Overall Response

| Overall | Overall (N=) |
|----------------------|--------------|
| Duration of response | |
| (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

4.7.5.1. FIGURE: WATERFALL PLOT. MAXIMUM % TOTAL CHANGE WITH BOR

- 4.7.5.2 FIGURE: WATERFALL PLOT. MAXIMUM % TOTAL CHANGE VS BOR
- 4.7.5.3 FIGURE: WATERFALL PLOT. MAXIMUM % TOTAL CHANGE VS PRIMARY LOCATION
- 4.7.5.4 FIGURE: WATERFALL PLOT. MAXIMUM % TOTAL CHANGE VS KI67
- 4.7.5.4 FIGURE: WATERFALL PLOT. MAXIMUM % TOTAL CHANGE VS DIFFERENTATION TUMOUR
- 4.7.5.2. FIGURE: SPIDER PLOT. MAXIMUM % TOTAL CHANGE

4.7.5.5 FIGURE: SPIDER PLOT. MAXIMUM % TOTAL CHANGE VS DIFFERENTIATION
4.7.5.6 FIGURE: SPIDER PLOT. MAXIMUM % TOTAL CHANGE VS BOR
4.7.5.7 FIGURE: SPIDER PLOT. MAXIMUM % TOTAL CHANGE VS CGA
4.7.5.8 FIGURE: SPIDER PLOT. MAXIMUM % TOTAL CHANGE VS NSE

# 4.8. OS STRATIFIED BY FACTORS OF INTEREST: DIFFERENTIATED/ K<sub>1</sub>67/ PRIMARY TUMOUR LOCATION / CGA / NSE

4.8.1.OS VS DIFFERENTIATION

Two groups are defined (as reported in eCRD): Well and Poorly differientated

Table 39: OS vs Differentiation: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|-----------------------|-----------------|--------|------|--------|
| Well differentiated | | | | |
| Poorly differentiated | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 40: OS vs Differentiation: Survival ratio estimation

| SG | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Well differentiated | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Poorly | | | | |
| differentiated | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.8.1.1. FIGURE: OS VS DIFFERENTIATION. KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.8.2.OS vs Kı67

Two groups are defined from the Ki67 values recorded at the eCRF: ≤ 55 and >55

Table 41: OS vs Ki67: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|----------|-----------------|--------|------|--------|
| Ki67<=55 | | | | |
| Ki67>55 | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 42: OS vs Ki67: Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Ki67<=55 | | | | |
| At 6 months | | | | |
| At 12 | | | | |
| months | | | | |
| Ki67>55 | | | | |
| At 6 months | | | | |
| At 12 | | | | |
| months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.8.2.1. FIGURE: OS VS KI67. KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.8.3.OS vs Location

Six groups are defined from the Location recorded at the eCRF: Esophagus/Gastric, Pancreas, Colon/Rectum, Duodenum/Ileum and Not specified/Others.

Table 43: OS vs Location: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|----------------------|-----------------|--------|------|--------|
| Duodenum/Ileum | | | | |
| Esophagus/Gastric | | | | |
| Pancreas | | | | |
| Colon/Rectum | | | | |
| Not specified/Others | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 44: OS vs Location Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Duodenum/lleum | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Esophagus/Gastri | | | | |
| С | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Pancreas | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Colon/Rectum | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Not | | | | |
| specified/Others | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.8.3.1. FIGURE: OS VS LOCATION. KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.8.4.OS vs CGA

Two groups are defined from the CGA recorded at the eCRF: CGA < 2\*ULN and CGA >= 2\*ULN.

Table 45: OS vs CGA: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|--------------|-----------------|--------|------|--------|
| CGA < 2*ULN | | | | |
| CGA >= 2*ULN | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 46: OS vs CGA Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| CGA < 2*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| CGA >= | | | | |
| 2*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.8.4.1. FIGURE: OS VS CGA KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.8.5.OS vs NSE

Two groups are defined from the Location recorded at the eCRF: NSE < 2\*ULN, NSE >= 2\*ULN

Table 47: OS vs NSE: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|--------------|-----------------|--------|------|--------|
| NSE < 2*ULN | | | | |
| NSE >= 2*ULN | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 48: OS vs NSE Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| NSE < 2*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| NSE >= | | | | |
| 2*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.8.5.1. FIGURE: OS VS NSE KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

# 4.9. PFS STRATIFIED BY FACTORS OF INTEREST: DIFFERENTIATED/ K<sub>1</sub>67/ PRIMARY TUMOUR LOCATION / CGA / ENOLASE

4.9.1.PFS vs DIFFERENTIATION

Two groups are defined (as reported in eCRD): Well and Poorly differentiated

Table 49: PFS vs Differentiation: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|-----------------------|-----------------|--------|------|--------|
| Well differentiated | | | | |
| Poorly differentiated | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 50: PFS vs Differentiation: Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Well differentiated | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Poorly | | | | |
| differentiated | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.9.1.1. FIGURE: PFS vs DIFFERENTIATION, KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.9.2.PFS vs Ki67

Two groups are defined from the Ki67 values recorded at the eCRF: <=55 and >55

Table 51: PFS vs Ki67: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|----------|-----------------|--------|------|--------|
| Ki67<=55 | | | | |
| Ki67>55 | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 52: PFS vs Ki67: Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Ki67<=55 | | | | |
| At 6 months | | | | |
| At 12 | | | | |
| months | | | | |
| Ki67>55 | | | | |
| At 6 months | | | | |
| At 12 | | | | |
| months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.9.2.1. FIGURE: PFS VS KI67. KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.9.3.PFS vs Location

Six groups are defined from the Location recorded at the eCRF: Esophagus/Gastric, Pancreas, Colon/Rectum, Duodenum/Ileum and Not specified/Others.

Table 53: PFS vs Location: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|----------------------|-----------------|--------|------|--------|
| Duodenum/Ileum | | | | |
| Esophagus/Gastric | | | | |
| Pancreas | | | | |
| Colon/Rectum | | | | |
| Not specified/Others | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 54: PFS vs Location Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Duodenum/lleum | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Esophagus/Gastri | | | | |
| С | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Pancreas | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Colon/Rectum | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| Not | | | | |
| specified/Others | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.9.3.1. FIGURE: PFS VS LOCATION. KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value= X

#### 4.9.4.PFS vs CGA 4.9.4.1. PFS vs CGA (2)

Two groups are defined from the CGA at the eCRF: CGA < 2\*ULN and CGA >= 2\*ULN.

Table 55: PFS vs CGA: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|--------------|-----------------|--------|------|--------|
| CGA < 2*ULN | | | | |
| CGA >= 2*ULN | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 56: PFS vs CGA: Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| CGA < 2*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| CGA >= | | | | |
| 2*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.9.4.2. FIGURE: PFS vs CGA KAPLAN MEIER GRAPH (2)

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.9.4.3. **PFS** vs **CGA** (3)

Two groups are defined from the CGA at the eCRF: CGA < 3·ULN and CGA >=  $3\cdot$  ULN.

Table 57: PFS vs CGA: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|--------------|-----------------|--------|------|--------|
| CGA < 3*ULN | | | | |
| CGA >= 3*ULN | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 58: PFS vs CGA: Survival ratio estimation

| SG | Events (%, total<br>N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| CGA < 3*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| CGA >= | | | | |
| 3*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.9.4.4. FIGURE: PFS vs CGA KAPLAN MEIER GRAPH (3)

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.9.4.5. PFS vs CGA (5)

Two groups are defined from the CGA at the eCRF: CGA < 5\*ULN and CGA >= 5\*ULN.

Table 59: PFS vs CGA: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|--------------|-----------------|--------|------|--------|
| CGA < 5*ULN | | | | |
| CGA >= 5*ULN | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 60: PFS vs CGA: Survival ratio estimation

| SG | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| CGA < 5*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| CGA >= | | | | |
| 5*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.9.4.6. FIGURE: PFS vs CGA KAPLAN MEIER GRAPH (5)

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

#### 4.9.5.PFS vs Enolase

Two groups are defined from the Enolase values: NSE < 2\*ULN and NSE >= 2\*ULN

Table 61: PFS vs Enolase: Median estimation

| | Median (months) | CI 95% | Mean | CI 95% |
|--------------|-----------------|--------|------|--------|
| NSE < 2*ULN | | | | |
| NSE >= 2*ULN | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

Table 62: PFS vs NSE: Survival ratio estimation

| SG | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| NSE < 2*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |
| NSE >= | | | | |
| 2*ULN | | | | |
| At 6 months | | | | |
| At 12 months | | | | |

<sup>&</sup>lt;sup>1</sup>Estimated using Kaplan-Meier product-limit method

4.9.5.1. FIGURE: PFS VS NSE KAPLAN MEIER GRAPH

<sup>&</sup>lt;sup>2</sup> Log rank test to compare categories: p-value=X

# 4.10.ORR STRATIFIED BY FACTORS OF INTEREST: DIFFERENTIATED/ K<sub>1</sub>67/ PRIMARY TUMOUR LOCATION / CGA / NSE

Table 63: ORR vs Differentiation

| | Well differentiated (N=) | Poorly differentiated (N=) | Total (N=) | p<br>value |
|---|---|---|---|---|
| Best Overall Response | | | | |
| PR | | | | |
| SD | | | | |
| PD | | | | |
| NE | | | | |
| Objective Response Rate | | | | _ |
| (ORR): CR or PR (BOR) | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

- 1. Fisher's Exact Test for Count Data
- 2. Pearson's Chi-squared test

Table 64: ORR vs Ki67

| | <=55 (N=) | >55 (N=) | Total (N=) | p<br>value |
|---|---|---|---|---|
| Best Overall Response | | | | |
| PR | | | | |
| SD | | | | |
| PD | | | | |
| NE | | | | |
| Objective Response Rate (ORR): CR or PR | | | | |
| (BOR) | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

- 1. Fisher's Exact Test for Count Data
- 2. Pearson's Chi-squared test

Table 65: ORR vs Location

| | Esophagus/<br>Gastric (N=) | Pancrea<br>s (N=) | Colon/Rectu<br>m (N=) | Duodenum/<br>Ileum (N=) | Not<br>specified/Others<br>(N=) | Total (N=) | p<br>value |
|---|---|---|---|---|---|---|---|
| BOR | | | | | | | |
| PR | | | | | | | |
| SD | | | | | | | |
| PD | | | | | | | |
| NE | | | | | | | |
| Objective Response Rate | | | | | | | |
| (ORR): CR or PR (BOR) | | | | | | | |
| Yes (CR/PR) | | | | | | | |
| No | | | | | | | |

1. Fisher's Exact Test for Count Data

Table 66: ORR vs Location

| | Colon/Rectum<br>(N=) | Others<br>(N=) | Total (N=) | p<br>value |
|---|---|---|---|---|
| Best Overall Response | | | | |
| PR | | | | |
| SD | | | | |
| PD | | | | |
| NE | | | | |
| Objective Response Rate (ORR): CR | | | | |
| or PR (BOR) | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

<sup>1.</sup> Fisher's Exact Test for Count Data

Table 67: ORR vs CGA

| | CGA < 2*ULN | CGA >= 2*ULN | Total (N=) | р |
|---|---|---|---|---|
| | (N=) | (N=) | ( , | value |
| Best Overall Response | | | | |
| PR | | | | |
| SD | | | | |
| PD | | | | |
| NE | | | | |
| Objective Response Rate (ORR): | | | | |
| CR or PR (BOR) | | | | |
| Yes (CR/PR) | | | | |
| No | | · | | • |
| | • | | ·- | |

- 1. Fisher's Exact Test for Count Data
- 2. Pearson's Chi-squared test

Table 68: ORR vs Enolase

| | NSE < 2*ULN<br>(N=) | NSE >= 2*ULN<br>(N=) | Total (N=) | p<br>value |
|---|---|---|---|---|
| Best Overall Response | | | | |
| PR | | | | |
| SD | | | | |
| PD | | | | |
| NE | | | | |
| Objective Response Rate (ORR): | | | | |
| CR or PR (BOR) | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

- 1. Fisher's Exact Test for Count Data
- 2. Pearson's Chi-squared test

## 4.10.1. MULTIVARIATE ANALYSIS OF PFS AND OS 4.10.1.1. Factors included in the multivariate analysis of the PFS (1)

Table 69: Factors included in the multivariate analysis of the PFS

| PD/Exitus | No (N=) | Yes (N=) | Total (N=) | p value |
|---|---|---|---|---|
| CGA <> 2 x ULN | , , | , , , | ` ' | • |
| Missing data | | | | |
| CGA < 2*ULN | | | | |
| CGA >= 2*ULN | | | | |
| Enolase <> 2 x ULN | | | | |
| Missing data | | | | _ |
| NSE < 2*ULN | | | | |
| NSE >= 2*ULN | | | | |
| Primary neuroendocrine tumour | | | | |
| Duodenum/Ileum | | | | |
| Esophagus/Gastric | | | | |
| Pancreas | | | | |
| Colon/Rectum | | | | |
| Not specified/Others | | | | |
| Differentiation | | | | |
| Well differentiated | | | | |
| Poorly differentiated | | | | |
| Ki-67 categorised | | | | |
| <=55 | | | | |
| >55 | | | | |
| ECOG | | | | |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| Gender | | | | |
| Female | | | | |
| Male | | | | |
| Age categorised by median (61 years) | | | | |
| <=61y | | | | |
| >61y | | | | |
| LDH | | | | |
| <= 2ULN | | | | |
| > 2ULN | | | | |

<sup>1.</sup> Fisher's Exact Test for Count Data

Table 70: PFS univariate and multivariate Cox model

| | | Univa | riate Co | x Regression | | | Multiva | ariate Co | x Regression | <u> </u> |
|---|---|---|---|---|---|---|---|---|---|---|
| Characteristic | N | Event N | HR <sup>1</sup> | 95% CI <sup>1</sup> | p-value | N | Event N | HR <sup>1</sup> | 95% CI <sup>1</sup> | p-value |
| CGA <> 2 x ULN | | | | | | | | | | |
| CGA < 2*ULN | | | | | | | | | | |
| CGA >= 2*ULN | | | | | | | | | | |
| Enolase <> 2 x ULN | | | | | | | | | | |
| NSE < 2*ULN | | | | | | | | | | |
| NSE >= 2*ULN | | | | | | | | | | |
| Primary neuroendocrine tumour | | | | | | | | | | |
| Duodenum/Ileum | | | | | | | | | | |
| Esophagus/Gastric | | | | | | | | | | |
| Pancreas | | | | | | | | | | |
| Colon/Rectum | | | | | | | | | | |
| Not specified/Others | | | | | | | | | | |
| Differentiation | | | | | | | | | | |
| Well differentiated | | | | | | | | | | |
| Poorly differentiated | | | | | | | | | | |
| Ki-67 categorised | | | | | | | | | | |
| <=55 | | | | | | | | | | |
| >55 | | | | | | | | | | |
| ECOG | | | | | | | | | | |
| 0 | | | | | | | | | | |
| 1 | | | | | | | | | | |
| 2 | | | | | | | | | | |
| Gender | | | | | | | | | | |
| Female | | | | | | | | | | |
| Male | | | | | | | | | | |
| Age categorised by median (61 years) | | | | | | | | | | |
| <=61y | | | | | | | | | | |
| >61y | | | | | | | | | | |
| LDH | | | | | | | | | | |
| <= 2ULN | | | | | | | | | | |

| | | Univa | riate Co | <b>Regression</b> | | Multivariate Cox Regression | | | | 1 |
|---|---|---|---|---|---|---|---|---|---|---|
| Characteristic | N | Event N | HR <sup>1</sup> | 95% CI <sup>1</sup> | p-value | N | Event N | HR <sup>1</sup> | 95% CI <sup>1</sup> | p-value |
| > 2ULN | | | | | | | | | | |

<sup>1</sup>HR = Hazard Ratio, CI = Confidence Interval

Note: Los p-valores marcados en negrita indican que el valor es estadísticamente significativo <0.05

Figure 3: Forest plot PFS Multivariate Cox Regression

### 4.10.1.2. FACTORS INCLUDED IN THE MULTIVARIATE ANALYSIS OF THE PFS (2)

Table 71: Factors included in the multivariate analysis of the PFS

| PD/Exitus | No (N=) | Yes (N=) | Total (N=) | p value |
|---|---|---|---|---|
| CGA <> 2 x ULN | | | | |
| Missing data | | | | |
| CGA < 2*ULN | | | | |
| CGA >= 2*ULN | | | | |
| Enolase <> 2 x ULN | | | | |
| Missing data | | | | |
| NSE < 2*ULN | | | | |
| NSE >= 2*ULN | | | | |
| Primary neuroendocrine tumour | | | | |
| Colon/Rectum | | | | |
| Others | | | | |
| Differentiation | | | | |
| Well differentiated | | | | |
| Poorly differentiated | | | | |
| Ki-67 categorised | | | | |
| <=55 | | | | |
| >55 | | | | |
| ECOG | | | | |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| Gender | | | | |
| Female | | | | |
| Male | | | | |
| Age categorised by median (x years) | | | | |
| <=xy | | | | |
| >xy | | | | |
| LDH | | | | |
| <= 2ULN | | | | |
| > 2ULN | | | | |

1. Fisher's Exact Test for Count Data

Table 72: PFS univariate and multivariate Cox model

| | | Univa | riate Co | <b>Regression</b> | | | Multiva | ariate Co | x Regression | n |
|---|---|---|---|---|---|---|---|---|---|---|
| Characteristic | N | Event N | HR <sup>1</sup> | 95% CI <sup>1</sup> | p-value | N | Event N | HR <sup>1</sup> | 95% Cl <sup>1</sup> | p-value |
| CGA <> 2 x ULN | | | | | | | | | | |
| CGA < 2*ULN | | | | | | | | | | |
| CGA >= 2*ULN | | | | | | | | | | |
| Enolase <> 2 x ULN | | | | | | | | | | |
| NSE < 2*ULN | | | | | | | | | | |
| NSE >= 2*ULN | | | | | | | | | | |
| Primary neuroendocrine tumour | | | | | | | | | | |
| Colon/Rectum | | | | | | | | | | |
| Others | | | | | | | | | | |
| Differentiation | | | | | | | | | | |
| Well differentiated | | | | | | | | | | |
| Poorly differentiated | | | | | | | | | | |
| Ki-67 categorised | | | | | | | | | | |
| <=55 | | | | | | | | | | |
| >55 | | | | | | | | | | |
| ECOG | | | | | | | | | | |
| 0 | | | | | | | | | | |
| 1 | | | | | | | | | | |
| 2 | | | | | | | | | | |
| Gender | | | | | | | | | | |
| Female | | | | | | | | | | |
| Male | | | | | | | | | | |
| Age categorised by median (x years) | | | | | | | | | | |
| <=61y | | | | | | | | | | |
| >61y | | | | | | | | | | |
| LDH | | | | | | | | | | |
| <= 2ULN | | | | | | | | | | |
| > 2ULN | | 4= | | 4:- OI - O | | | | | | |

<sup>1</sup>HR = Hazard Ratio, CI = Confidence Interval

Note: Los p-valores marcados en negrita indican que el valor es estadísticamente significativo <0.05

Figure 4: Forest plot PFS Multivariate Cox Regression

### 4.10.1.3. FACTORS INCLUDED IN THE MULTIVARIATE ANALYSIS OF THE OS (1)

Table 73: Factors included in the multivariate analysis of the OS

| OS | Alive (N=) | Death (N=) | Total (N=) | p value |
|---|---|---|---|---|
| CGA <> 2 x ULN | | · | | · |
| Missing data | | | | |
| CGA < 2*ULN | | | | |
| CGA >= 2*ULN | | | | |
| Enolase <> 2 x ULN | | | | |
| Missing data | | | | |
| NSE < 2*ULN | | | | |
| NSE >= 2*ULN | | | | |
| Primary neuroendocrine tumour | | | | |
| Duodenum/Ileum | | | | |
| Esophagus/Gastric | | | | |
| Pancreas | | | | |
| Colon/Rectum | | | | |
| Not specified/Others | | | | |
| Differentiation | | | | |
| Well differentiated | | | | |
| Poorly differentiated | | | | |
| Ki-67 categorised | | | | |
| <=55 | | | | |
| >55 | | | | |
| ECOG | | | | |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| Gender | | | | |
| Female | | | | |
| Male | | | | |
| Age categorised by median (x years) | | | | |
| <=61y | | | | |
| >61y | | | | |
| LDH | | | | |

| OS | Alive (N=) | Death (N=) | Total (N=) | p value |
|---------|------------|------------|------------|---------|
| <= 2ULN | | | | _ |
| > 2ULN | | | | |

- 1. Fisher's Exact Test for Count Data
- 2. Pearson's Chi-squared test

Table 74: OS univariate and multivariate Cox model

| | | Univ | ariate Cox | Regression | | | Multi | variate Co | x Regression | |
|---|---|---|---|---|---|---|---|---|---|---|
| Characteristic | N | Event<br>N | HR¹ | 95% CI <sup>1</sup> | p-valu<br>e | N | Event<br>N | HR¹ | 95% CI <sup>1</sup> | p-valu<br>e |
| CGA <> 2 x ULN | | | | | | | | | | |
| CGA < 2*ULN | | | | | | | | | | |
| CGA >= 2*ULN | | | | | | | | | | |
| Enolase <> 2 x ULN | | | | | | | | | | |
| NSE < 2*ULN | | | | | | | | | | |
| NSE >= 2*ULN | | | | | | | | | | |
| Primary neuroendocrine tumour | | | | | | | | | | |
| Duodenum/lleum | | | | | | | | | | |
| Esophagus/Gastric | | | | | | | | | | |
| Pancreas | | | | | | | | | | |
| Colon/Rectum | | | | | | | | | | |
| Not specified/Others | | | | | | | | | | |
| Differentiation | | | | | | | | | | |
| Well differentiated | | | | | | | | | | |
| Poorly differentiated | | | | | | | | | | |
| Ki-67 categorised | | | | | | | | | | |
| <=55 | | | | | | | | | | |
| >55 | | | | | | | | | | |
| ECOG | | | | | | | | | | |
| 0 | | | | | | | | | | |
| 1 | | | | | | | | | | |
| 2 | | | | | | | | | | |
| Gender | | | | | | | | | | |
| Female | | | | | | | | | | |
| Male | | | | | | | | | | |
| Age categorised by median (x years) | | | | | | | | | | |
| <=61y | | | | | | | | | | |
| >61y | | | | | | | | | | |
| LDH | | | | | | | | | | |

| | Univariate Cox Regression | | | | | Multivariate Cox Regression | | | |
|---|---|---|---|---|---|---|---|---|---|
| Characteristic | l Event<br>N | HR <sup>1</sup> | 95% CI <sup>1</sup> | p-valu<br>e | N | Event<br>N | HR <sup>1</sup> | 95% CI <sup>1</sup> | p-valu<br>e |
| <= 2ULN | | | | | | | | | |
| > 2ULN | | | | | | | | | |

<sup>1</sup>HR = Hazard Ratio, CI = Confidence Interval

Note: Los p-valores marcados en negrita indican que el valor es estadísticamente significativo <0.05

Figure 5: Forest plot OS Multivariate Cox Regression

#### 4.10.1.4. FACTORS INCLUDED IN THE MULTIVARIATE ANALYSIS OF THE OS (2)

Table 75: Factors included in the multivariate analysis of the OS

| OS | Alive (N=) | Death (N=) | Total (N=) | p value |
|---|---|---|---|---|
| CGA <> 2 x ULN | | | | |
| Missing data | | | | |
| CGA < 2*ULN | | | | |
| CGA >= 2*ULN | | | | |
| Enolase <> 2 x ULN | | | | |
| Missing data | | | | |
| NSE < 2*ULN | | | | |
| NSE >= 2*ULN | | | | |
| Primary neuroendocrine tumour | | | | |
| Colon/Rectum | | | | |
| Others | | | | |
| Differentiation | | | | |
| Well differentiated | | | | |
| Poorly differentiated | | | | |
| Ki-67 categorised | | | | |
| <=55 | | | | |
| >55 | | | | |
| ECOG | | | | |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| Gender | | | | |
| Female | | | | |
| Male | | | | |
| Age categorised by median (61 years) | | | | |
| <=61y | | | | |
| >61y | | | | |
| LDH | | | | |
| <= 2ULN | | | | |
| > 2ULN | | | | |

- 1. Fisher's Exact Test for Count Data
- 2. Pearson's Chi-squared test

Table 76: OS univariate and multivariate Cox model

| | | Univa | riate Co | x Regression | | | Multiva | ariate Co | x Regression | 1 |
|---|---|---|---|---|---|---|---|---|---|---|
| Characteristic | N | Event N | $HR^1$ | 95% CI <sup>1</sup> | p-value | N | Event N | $HR^1$ | 95% CI <sup>1</sup> | p-value |
| CGA <> 2 x ULN | | | | | | | | | | |
| CGA < 2*ULN | | | | | | | | | | |
| CGA >= 2*ULN | | | | | | | | | | |
| Enolase <> 2 x ULN | | | | | | | | | | |
| NSE < 2*ULN | | | | | | | | | | |
| NSE >= 2*ULN | | | | | | | | | | |
| Primary neuroendocrine tumour | | | | | | | | | | |
| Colon/Rectum | | | | | | | | | | |
| Others | | | | | | | | | | |
| Differentiation | | | | | | | | | | |
| Well differentiated | | | | | | | | | | |
| Poorly differentiated | | | | | | | | | | |
| Ki-67 categorised | | | | | | | | | | |
| <=55 | | | | | | | | | | |
| >55 | | | | | | | | | | |
| ECOG | | | | | | | | | | |
| 0 | | | | | | | | | | |
| 1 | | | | | | | | | | |
| 2 | | | | | | | | | | |
| Gender | | | | | | | | | | |
| Female | | | | | | | | | | |
| Male | | | | | | | | | | |
| Age categorised by median (61 years) | | | | | | | | | | |
| <=61y | | | | | | | | | | |
| >61y | | | | | | | | | | |
| LDH | | | | | | | | | | |
| <= 2ULN | | | | | | | | | | |
| > 2ULN | | | | | | | | | | |

<sup>1</sup>HR = Hazard Ratio, CI = Confidence Interval

 $^{ ext{Note:}}$  Los p-valores marcados en negrita indican que el valor es estadísticamente significativo <0.05

Figure 6: Forest plot OS Multivariate Cox Regression

## 5. SAFETY ANALYSIS

Table 77: Overall safety

| | Induction (N=) | Maintenance (N=) | General (N=) |
|---|---|---|---|
| Any AE | | | |
| Yes | | | |
| No | | | |
| AE grade >=3 | | | |
| Yes | | | |
| No | | | |
| Toxicity: AE related to any treatment | | | |
| Yes | | | |
| No | | | |
| Toxicity: AE related to nivolumab | | | |
| Yes | | | |
| No | | | |
| Toxicity: AE related to carboplatin | | | |
| Yes | | | |
| No | | | |
| Toxicity: AE related to etoposide | | | |
| Yes | | | |
| No | | | |
| Toxicity: AE related to all treatments (induction) | | | |
| Yes | | | |
| No | | | |
| Toxicity grade >=3 | | | |
| Yes | | | |
| No | | | |
| Toxicity related to nivolumab grade >=3 | | | |
| Yes | | | |
| No | | | |
| Toxicity related to carboplatin grade >=3 | | | |
| Yes | | | |
| No | | | |
| Toxicity related to etoposide grade >=3 | | | |
| Yes | | | |
| No | | | |
| Toxicity related to all treatments grade >=3 | | | |
| (induction) | | | |
| Yes | | | |
| No | | | |
| SAE | | | |
| Yes | | | |
| No | | | |

### 5.1. INDUCTION

Table 78: Most frequent Toxicity with 5% threshold (induction)

| ige (%) |
|---------|

Table 79: Grade of most frequent toxicities with 5% threshold overall (induction)

| Toxicity | No | G-UK | G-1 | G-2 | G-3 | G-4 | G-5 |
|----------|----|------|-----|-----|-----|-----|-----|

Table 80: List of toxicities grade >= 3 in all patients (induction)

| Patient Number | AE CTCAE | AE Grade | AE Related to |
|----------------|----------|----------|---------------|

Table 81: Most frequent AEs with 5% threshold (induction)

Table 82: Grade of most frequent AEs with 5% threshold overall (induction)

| AE | No | G-UK | G-1 | G-2 | G-3 | G-4 | G-5 |
|----|----|------|-----|-----|-----|-----|-----|

Table 83: List of all SAEs (induction)

| Patient<br>Number | AE CTCAE | AE CTCAE AE<br>Other Grad | e AE Start Date AE Stop Date Related | AE Intensity | AE Related to |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

Table 84: List of all toxicities (induction)

| Patient<br>Number | AE CTCAE | AE CTCAE<br>Other | AE<br>Grade | AE Start<br>Date | AE Stop<br>Date | AE<br>SAE | AE<br>Intensity | AE Related to |
|---|---|---|---|---|---|---|---|---|

#### 5.2. MAINTENANCE

Table 85: Most frequent Toxicity with 5% threshold (maintenance)

| Toxicity | Frequency | Percentage (%) |
|----------|-----------|----------------|

Table 86: Grade of most frequent toxicities with 5% threshold overall (maintenance)

| Toxicity | No | G-UK | G-1 | G-2 | G-3 | G-4 | G-5 |
|----------|----|------|-----|-----|-----|-----|-----|

Table 87: List of toxicities grade >=3 in all patients (maintenance)

| Patient Number | AE CTCAE | AE Grade | AE Related to |
|----------------|----------|----------|---------------|

Table 88: Most frequent AEs with 5% threshold (maintenance)



Table 89: Grade of most frequent AEs with 5% threshold overall (maintenance)

| AE | No | G-UK | G-1 | G-2 | G-3 | G-4 | G-5 |
|----|----|------|-----|-----|-----|-----|-----|

Table 90: List of all SAEs (maintenance)

| Patient<br>Number | AE CTCAE | AE CTCAE<br>Other | AE<br>Grade | AE Start<br>Date | AE Stop<br>Date | AE<br>Related | AE Intensity | AE<br>Related<br>to |
|---|---|---|---|---|---|---|---|---|

Table 91: List of all toxicities (maintenance)

| Patient<br>Number | AE CTCAE | AE CTCAE Other Grade | AE Start<br>Date | AE Stop<br>Date | AE<br>SAE | AE Intensity | AE Related to |
|---|---|---|---|---|---|---|---|

#### 5.3. GENERAL

Table 92: Most frequent Toxicity with 5% threshold

| Frequency | Percentage (%) |
|-----------|----------------|
| | Frequency |

Table 93: Grade of most frequent toxicities with 5% threshold overall

| Toxicity | No | G-UK | G-1 | G-2 | G-3 | G-4 | G-5 |
|----------|----|------|-----|-----|-----|-----|-----|

Table 94: List of toxicities grade >=3 in all patients

| Patient Number | AE CTCAE | AE Grade | AE Related to |
|----------------|----------|----------|---------------|

Table 95: Most frequent AEs with 5% threshold

| AE | Frequency | Percentage (%) |
|----|-----------|----------------|

Table 96: Grade of most frequent AEs with 5% threshold overall

| AE | No | G-UK | G-1 | G-2 | G-3 | G-4 | G-5 |
|----|----|------|-----|-----|-----|-----|-----|

Table 97: List of all SAEs

| Patient<br>Number | AE CTCAE | AE CTCAE<br>Other | AE<br>Grade | AE Start Date AE Stop Date AE Related AE Intensity AE Related to |
|---|---|---|---|---|

Table 98: List of all toxicities

| Patient<br>Number | AE CTCAE | AE CTCAE Other Grade | AE Start<br>Date | AE Stop<br>Date | AE<br>SAE | AE Intensity | AE Related to |
|---|---|---|---|---|---|---|---|